CLINICAL TRIAL: NCT03210519
Title: A Randomized, Double-blind, Placebo-controlled Trial to Evaluate the Efficacy of Eleutherococcus Senticosus for Anti-inflammation and Improvement of Erythropoietin Hyporesponsiveness in Subjects Under Renal Dialysis
Brief Title: To Evaluate the Efficacy of Eleutherococcus Senticosus for Subjects Under Renal Dialysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chung Shan Medical University (Other)
Responsible Party: Principal Investigator, Nae-Cherng Yang, Associate Professor, Chung Shan Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CS15036
Record Dates: First submitted 2017-07-03; First posted 2017-07-07 (Actual); Results first posted 2020-05-06 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Renal Dialysis
MeSH Terms: interventions — Siberian ginseng root

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Eleutherococcus senticosus (Experimental): Acanthopanax senticosus-mono formula (30mg/vial) and Fructus Ziziphi Jujube concentrated juice15ml/vial
  Interventions: Dietary Supplement: Eleutherococcus senticosus
- Placebo (Placebo Comparator): Fructus Ziziphi Jujube concentrated juice15ml/vial
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Eleutherococcus senticosus — taken orally once/day for 90 days
  Arms: Eleutherococcus senticosus
Other: Placebo — taken orally once/day for 90 days
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled, parallel comparison trial to evaluate the efficacy and safety of Eleutherococcus Senticosus taken orally by patients under regular dialysis. Eligible subjects with written consent were randomized into one of the two groups: A. Acanthopanax senticosus (30mg/vial); B. Placebo. After 2-4 weeks of run-in period, the study subjects were asked to take the investigational products orally for 90 days in order to evaluate the effects of oral Eleutherococcus Senticosus liquid on the markers of inflammation, anemia, and safety, and to compare the efficacy among oral Acanthopanax senticosus and placebo.

ELIGIBILITY:
Inclusion Criteria:

* Under regular dialysis for at least 3 months
* Hemoglobin (Hb) <11 g/L after regular Erythropoietin (EPO) treatment
* Subjects with written informed consent form

Exclusion Criteria:

* Use of steroid or high dose of antiplatelet drug (e.g. Aspirin >300mg) within one month
* Had surgery, myocardial infarction, or tumor within 12 weeks
* Currently use of antibiotic treatment for acute infection
* Pregnant women
* Reticulocyte>40 x 10^9
* Anemia (ferritin <100ng/mL and Transferrin Saturation (TSAT) <20%)
* Urea reduction ratio <65% or single pool Kt/V < 1.0 (hemodialysis patients) or total weekly Kt/V<1.7 (peritoneal dialysis patients)
* Sudden change of eating habit within one month
* Expected life less than six months or with unstable medical conditions
* Known history of allergic reaction to the investigational products
* With acute diseases and judged by the investigator to be ineligible to participate
* Received melatonin, androgen therapy or blood transfusion within two months
* Received any trial medications within 30 days

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2015-12-09 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nae-Cherng Yang, Ph. D., Principal Investigator — Chun Shan Medical University

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Eleutherococcus Senticosus: Participants first received screening tests for up to 30 days. Eligible subjects were then given the investigational products (Acanthopanax senticosus-mono formula 30mg/vial and Fructus Ziziphi Jujube concentrated juice15ml/vial) to be taken orally once/day for 90 days. Patients with hyperacidity and gastroesophageal reflux were recommended to take it after meals.
- Placebo: Participants first received screening tests for up to 30 days. Eligible subjects were then given the investigational products (Fructus Ziziphi Jujube concentrated juice15ml/vial) to be taken orally once/day for 90 days. Patients with hyperacidity and gastroesophageal reflux were recommended to take it after meals.
Period: Overall Study
Arm/Group | Eleutherococcus Senticosus | Placebo
Started | 11 | 10
Completed | 9 | 10
Not Completed | 2 | 0
Not completed — Adverse Event | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Eleutherococcus Senticosus | Placebo | Total
Number analyzed (Participants) | 11 | 10 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (13.1) | 55.8 (11.3) | 60.1 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 11
  Male | 6 | 4 | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Taiwan | 11 | 10 | 21

OUTCOME MEASURES:

1. Primary Outcome: Erythropoietin (EPO)
Description: value at 3 months minus value at baseline reported
Time Frame: baseline and 3 months
Measure: Mean (Standard Deviation); unit: u/mth
Arm/Group | Eleutherococcus Senticosus | Placebo
Number analyzed (Participants) | 9 | 10
u/mth | -6000.0 (5916.5) | -1714.3 (6264.1)

2. Primary Outcome: Hemoglobin (Hb)
Description: value at 3 months minus value at baseline reported
Time Frame: baseline and 3 months
Measure: Mean (Standard Deviation); unit: gm/dl
Arm/Group | Eleutherococcus Senticosus | Placebo
Number analyzed (Participants) | 9 | 10
gm/dl | 1.0 (1.1) | -0.1 (0.8)

3. Secondary Outcome: Red Blood Cell (RBC)
Description: value at 3 months minus value at baseline reported
Time Frame: baseline and 3 months
Measure: Mean (Standard Deviation); unit: 10^4 cells/ul
Arm/Group | Eleutherococcus Senticosus | Placebo
Number analyzed (Participants) | 9 | 10
10^4 cells/ul | 25.1 (35.6) | -7.8 (28.7)

4. Secondary Outcome: Hematocrit (Hct)
Description: value at 3 months minus value at baseline reported
Time Frame: baseline and 3 months
Measure: Mean (Standard Deviation); unit: vol% RBC in blood
Arm/Group | Eleutherococcus Senticosus | Placebo
Number analyzed (Participants) | 9 | 10
vol% RBC in blood | 2.5 (3.2) | -0.3 (2.6)

5. Secondary Outcome: Mean Corpuscular Hemoglobin Concentration (MCHC)
Description: value at 3 months minus value at baseline reported
Time Frame: baseline and 3 months
Measure: Mean (Standard Deviation); unit: g/dl
Arm/Group | Eleutherococcus Senticosus | Placebo
Number analyzed (Participants) | 9 | 10
g/dl | -0.5 (0.3) | -0.3 (1.0)

6. Secondary Outcome: Mean Corpuscular Volume (MCV)
Description: value at 3 months minus value at baseline reported
Time Frame: baseline and 3 months
Measure: Mean (Standard Deviation); unit: fl
Arm/Group | Eleutherococcus Senticosus | Placebo
Number analyzed (Participants) | 9 | 10
fl | 1.3 (3.0) | 1.7 (2.2)

7. Secondary Outcome: Mean Corpuscular Hemoglobin (MCH)
Description: value at 3 months minus value at baseline reported
Time Frame: baseline and 3 months
Measure: Mean (Standard Deviation); unit: Pg
Arm/Group | Eleutherococcus Senticosus | Placebo
Number analyzed (Participants) | 9 | 10
Pg | 0.0 (1.1) | 0.3 (0.7)

8. Secondary Outcome: Intact Parathyroid Hormone (iPTH)
Description: value at 3 months minus value at baseline reported
Time Frame: baseline and 3 months
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Eleutherococcus Senticosus | Placebo
Number analyzed (Participants) | 9 | 10
pg/ml | 28.6 (240.5) | -97.9 (149.3)

9. Secondary Outcome: Tumor Necrosis Factor - Alpha (TNF-alpha)
Description: value at 3 months minus value at baseline reported
Time Frame: baseline and 3 months
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Eleutherococcus Senticosus | Placebo
Number analyzed (Participants) | 9 | 10
pg/ml | -17.2 (16.1) | -14.9 (19.6)

10. Secondary Outcome: Interleukin 6 (IL-6)
Description: value at 3 months minus value at baseline reported
Time Frame: baseline and 3 months
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Eleutherococcus Senticosus | Placebo
Number analyzed (Participants) | 9 | 10
pg/ml | -20.3 (28.7) | -0.7 (41.2)

ADVERSE EVENTS:
Time Frame: 1 and 3 months
Description: Vital signs and patients' self-evaluation of their tolerance and physical improvement was assessed by a structured patient questionnaire administered at months 1 and 3
Arm/Group | Eleutherococcus Senticosus | Placebo
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/10
Other Adverse Events (participants affected / at risk) | 2/11 | 0/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Eleutherococcus Senticosus (N=11) | Placebo (N=10)
Subjects complained uncomfortable (Gastrointestinal disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-06-05): https://cdn.clinicaltrials.gov/large-docs/19/NCT03210519/Prot_SAP_000.pdf